CLINICAL TRIAL: NCT07396948
Title: The Effectiveness of Two Physiotherapy Protocols in the Treatment of Patellofemoral Pain Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KB/134/2025
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Patellofemoral Disorder
Keywords: patellofemoral pain syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- training protocol (Placebo Comparator): Training protocol with three exercises
  Interventions: Other: training protocol
- medial patellar mobilization (Active Comparator)
  Interventions: Other: medial patellar mobilization
- quadriceps muscle stretching (Active Comparator)
  Interventions: Other: quadriceps muscle stretching

INTERVENTIONS:
Other: medial patellar mobilization — Patellar mobilization was carried out three times for 60 seconds each session [19]. The technique was performed by placing the therapist's thumbs on the lateral edge of the patella allowing a patellar glide in the medial and slightly caudal direction. The aim of this technique was to stretch the lateral patellar retinaculum
  Arms: medial patellar mobilization
Other: quadriceps muscle stretching — In order to perform this technique the patient was positioned prone on a treatment table (Figure 6). The non-stretched limb remained on the ground, flexed at the hip and knee. Moving this limb forward ensured proper aligment of the lumbar spine, while elevating the heel and placing it on the therapist's foot reduced tension in the hamstring group. Proper execution of the technique could be performed when the pelvis was aligned parallel to the surface, keeping the trunk and thigh of the stretched limb in one line. The therapist grasped by ipsilateral hand the distal third of the patient's lower leg and pulled the heel toward the buttock while by the contralateral hand stabilized the pelvis. The static position of stretching was maintained for 30 seconds in every repetition.
  Arms: quadriceps muscle stretching
Other: training protocol — The training protocol included the following exercise:
  glute bridges, half squat, rear lunges, side walk with elastic band
  Arms: training protocol

SUMMARY:
Patellofemoral pain syndrome (PFPS) is one of the most common causes of anterior knee pain in young and active individuals. PFPS is characterized by anterior knee pain. The treatment of choice is conservative management. However, there is still lack of widely accepted physiotherapeutic strategies aimed at alleviating patellofemoral pain. The outcomes of conservative treatment remain unsatisfactory. Therefore, the aim of this study was to compare the effectiveness of two physiotherapy protocols based on manual therapy and muscle training in the treatment of patellofemoral pain

ELIGIBILITY:
Inclusion Criteria: anterior knee pain (unilateral or bilateral) lasting at least one month -

Exclusion Criteria: previous knee injuries or surgeries, systemic diseases, patellar dislocation or subluxation, patellar maltracking, ligamentous laxity, patellar tendon pathologies, spinal pain, other abnormalities such as leg length discrepancy >2 cm, patients treated pharmacologically, with physiotherapy, or acupuncture in the knee area within the past 30 days

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-01-22 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
AKPS score | 6 weeks
VAS scale | 6 weeks